CLINICAL TRIAL: NCT01128803
Title: Phase I/II Multicenter: Immunotherapy of Hepatocellular Carcinoma by Induction of Anti-alpha Fetoprotein Response
Brief Title: Immunotherapy of Hepatocellular Carcinoma by Induction of Anti-alpha Fetoprotein Response
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06/9-P
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; immunotherapy; alpha foetoprotein; dendritic cells
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: injection of the cell therapy product — Between D-15 and D-30: Cytapheresis D0: 1st injection of the cell therapy product D21: 2nd injection of the cell therapy product D42: 3rd injection of the cell therapy product and 1 injection of dendritic cells not loaded D45: cutaneous biopsies if induration > 2mm

SUMMARY:
The secretion by tumor cells of alpha fetoprotein (AFP) was observed in 50 to 60% of hepatocellular carcinoma. The AFP can be used as a marker for tumor recurrence after treatment and may be considered as a tumor antigen specific for hepatocellular carcinoma.The aim of the project is to use the alpha fetoprotein (AFP) as a tumor antigen and to propose an approach of immunotherapy for hepatocellular carcinoma based on the injection of autologous dendritic cells loaded with specific peptides of AFP.

ELIGIBILITY:
Pre-inclusion Criteria :

* Adults (men or women) aged between 18 and 80 years
* Patients affiliated to a social security reimbursement system
* Signed informed consent
* Hepatocellular carcinoma
* At least one dosage with Alpha-foeto-protein ≥ 40 ng/ml
* Patient already treated with chemoembolization, percutaneous destruction (alcohol or radiofrequency), surgery or Sorafenib.

Inclusion Criteria:

* Negative test for pregnancy or effective contraception
* Patient HIV-, Hep B-, Hep C-, HTLV1 and 2-, Syphilis-
* HLA A 0201 group

Exclusion Criteria:

* Life expectancy < 3 months
* Pregnancy or breast-feeding
* Severe auto-immune disease
* Another malignant tumor except if considered as cured since more than 5 years
* History of uncontrolled psychiatric condition
* Risk factors of Creutzfeldt Jacobs disease
* Decompensated cirrhosis(ascites or Child-Pugh score greater than 8)
* Hepatic transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 days after each injection
  The main aim of this study is to test the absence of toxicity of the injection of autologist dendritic cells loaded with specific peptides of the AFP, for patients with hepatocellular carcinoma and already treated.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 weeks after the last injection
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 months after the last injection

SECONDARY OUTCOMES:
Analysis of T lymphocytes | before each injection
  The secondary aim of the study is to evaluate the anti-AFP immunizing response among patients who received the treatment
Analysis of T lymphocytes | 3 weeks after the last injection
Analysis of T lymphocytes | 3 months after the last injection

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme GOURNAY, Dr, Principal Investigator — Nantes University Hospital
Locations (4):
- France (4):
  - University Hospital of Angers, Angers
  - CHD La Roche-sur-Yon, La Roche-sur-Yon
  - Nantes University Hospital, Nantes
  - CH Saint Nazaire, Saint-Nazaire